CLINICAL TRIAL: NCT06196970
Title: Effects of Pilates and Burpees Exercises on Core Strengthening and Dynamic Balance in Cricket Players
Brief Title: Effects of Pilates and Burpees Exercises in Core Strengthening and Dynamic Balance.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0458
Record Dates: First submitted 2023-11-09; First posted 2024-01-09 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Sports Physical Therapy
Keywords: Pilates exercise; Burpees exercises; Core strengthening; Dynamic balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline warmup along with Pilate exercises (Experimental): Pilate exercises: Group A perform Pilates exercises for 6 weeks. In the initial stage of training Pilates exercises with lo intensity then we proceeded gradually with high intensity. Pilates was performed for core strengthening and dynamic balance Pelvic curl, The hundred, Side plank with 4-5 rep, 30 sec hold and 3 sets with each exercise.
  Interventions: Other: Pilate exercises
- : Baseline physical therapy treatment along with burpees exercises (Experimental): Burpees Exercises: Group B perform Burpees exercises for 6 weeks. In initial weeks of training Burpees exercises with low intensity then we proceeded gradually with high intensity exercises. Burpees was performed for core strengthening and dynamic balance .10 to 15 repetition ,3 sets with rest interval of 10 sec after each set of exercises
  Interventions: Other: Burpees exercises

INTERVENTIONS:
Other: Pilate exercises — After 10 minutes of warmup excercises, participatants perform pilates exercises, Pelvic curl : 45 seconds hold The Hundred : 45 seconds hold Bird Dog : 45 seconds hold Side plank : 45 seconds hold Frequency 3 days a week intensity 45 minutes hold a pose. Time will be 10 to 15 minutes.
  Arms: Baseline warmup along with Pilate exercises
Other: Burpees exercises — After 10 minutes of warmup excercises, participatants perform burppes excercises.
  1. Stand straight with your feet shoulder-width apart.
  2. Squat and place your hands in front of your feet.
  3. Jump back until your legs are fully extended and your body is in plank position.
  4. Do a push up, jump forward, and then push through the heels to return to the starting position.
  5. Repeat until the set is complete. Frequency 3 days a week .Time 10 to 15 minutes with 10 reputation , 3 sets. Rest internal will be 10 seconds after each set.
  Arms: : Baseline physical therapy treatment along with burpees exercises

SUMMARY:
This study will be a randomized clinical trial will be conducted in Ayub national park cricket club Sample size will be 48 to evaluate the effects of Pilates and Burpees exercises training among cricket players with an age range of 16-24 years. Non probability convenient sampling technique would be used. Participants will be randomly assigned to 2 groups. Group A will include participants who received Pilates exercises training (6 weeks) along with the warm up. Group B participant who will receive burpees exercise training (6 weeks) and warm up. Outcomes of both trainings are the effects on core strengthening and dynamic balance on players in A group and the B group. Post interventional assessment was done via Star excursion balance test, prone bridge test and 1 minute sit-up test. Data will be collected at baseline and 6 weeks. Data will be analyzed by SPSS version 25

DETAILED DESCRIPTION:
Cricket is a most popular sport played throughout the world. It is played in three common formats depending on the duration of the game, firstly a Test match is played over 4-5 day's with around 90 overs per day Secondly One day match is shorter with 50 over on each side and the Last one is T-Twenty match much shorter with 20 over on each side. As each format places different physical demands on the players the require an extensive combination of tactics, skills and physical fitness in the form of strength, flexibility and balance. In our study we can focus on the basic core strengthening which is essential for physical fitness and better performance in the game. Primary the aim of this study is to evaluate the comparative effects of Pilates and Burpees exercises of core strengthening and dynamic stability of body in young cricket players

ELIGIBILITY:
Inclusion Criteria:

* Partipant should be a cricket player.
* Individual with age group of 16-24 years.
* Only male players without any history of fracture

Exclusion Criteria:

* Player who recieved any type of physical therapy session during last 2 months.
* Any type of soft tissue injury reported.
* Any type of deformity.
* Past history of surgical procedures.

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Star excursion balance test: | Pre and 6 week post interventional
  Star Excursion Balance test is a dynamic test required for proprioception along with strength and flexibility. It is a measure of dynamic balance providing challenge to athletes and physically active individual
One min situp test: | Pre and 6 week post interventional
  Abdominal muscle strength and endurance is important for core stability and back support. This sit-up test measures the strength and endurance of the abdominals and hip-flexor muscles
Prone bridges test: | Pre and 6 week post interventional
  The prone bridge provides an indication of core abdominal strength.Prior to undertaking this test a member of the Health Promotion Unit will explain the test protocol and provide a demonstration to the group of Applicants

CONTACTS AND LOCATIONS:
Overall Officials: Imran Ghafoor, PhD, Principal Investigator — Riphah International University
Locations (1):
- Abdul Rahman Hashmi, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 2. Kamatchi K, Arun B, Tharani G, Yuvarani G, Vaishnavi G, Kaviraja NJB. Effects of swiss ball exercise and pilates exercise on core muscle strengthening in college cricketers. 2020;40(3):377-80.
- [Background] Pote L, Christie CJ. Strength and Conditioning Practices of University and High School Level Cricket Coaches: A South African Context. J Strength Cond Res. 2016 Dec;30(12):3464-3470. doi: 10.1519/JSC.0000000000001432. PMID 27075640
- [Background] 4. Bandyopadhyay KJSiS. Pakistani Cricket at Crossroads: An Outsider's Perspective. 2007;10(1):101-19.
- [Background] Cicchese JM, Evans S, Hult C, Joslyn LR, Wessler T, Millar JA, Marino S, Cilfone NA, Mattila JT, Linderman JJ, Kirschner DE. Dynamic balance of pro- and anti-inflammatory signals controls disease and limits pathology. Immunol Rev. 2018 Sep;285(1):147-167. doi: 10.1111/imr.12671. PMID 30129209
- [Background] 6. Manna C, Thander AJI. A comparative study of suryanamaskar and dynamic stretching on fast bowling performance in cricket. 2021;7(5):20-3.
- [Background] 7. Peng S, Li L, Wu HB, Madhavi S, Lou XWJAEM. Controlled growth of NiMoO4 nanosheet and nanorod arrays on various conductive substrates as advanced electrodes for asymmetric supercapacitors. 2015;5(2):1401172.
- [Background] Huxel Bliven KC, Anderson BE. Core stability training for injury prevention. Sports Health. 2013 Nov;5(6):514-22. doi: 10.1177/1941738113481200. PMID 24427426
- [Background] 9. Goel A, Pramanik AJCEP. Effect of post-activation potentiation using core activation on isometric core strength and countermovement jump variables in university male recreational athletes. 2022;18(5):375-84.